CLINICAL TRIAL: NCT00108433
Title: Linezolid vs Vancomycin/Cefazolin in the Treatment of Hemodialysis Patients With Catheter-Related Gram-Positive Bloodstream Infections
Brief Title: Linezolid in the Treatment of Hemodialysis Patients With Catheter-Related Gram-Positive Bloodstream Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5951105
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-06

CONDITIONS: Bacteremia; Gram-Positive Bacterial Infections
MeSH Terms: conditions — Bacteremia; Gram-Positive Bacterial Infections | interventions — Vancomycin

INTERVENTIONS:
Drug: Cefazolin IV
Drug: Linezolid IV
Drug: Vancomycin (IV)

SUMMARY:
This study will treat hemodialysis patients who have a central catheter that is thought to be infected with a specific bacteria (Gram positive bacteria).

DETAILED DESCRIPTION:
Pfizer suspended enrollment on 21 August 2006 as a precautionary measure in light of the mortality imbalance seen in a similar study, and terminated the study on April 6, 2007 due to factors affecting the timeline to completion, such as slow enrollment and inclusion of sufficient evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, a patient must provide informed consent and must meet all of the following criteria. No study procedures, including any baseline tests, should be performed until the patient (or parent/legally acceptable representative, if appropriate) legally signs the informed consent form.
* Male or female, 18 years of age or older and >= 40 kg body weight
* End-stage renal disease patients on hemodialysis with: A) Signs and symptoms of a localized catheter-related infection (eg tenderness and/or pain, erythema, swelling, purulent exudates within 2 cm of entry site); OR B) A body temperature of >= 38.0 C or < 36.0 C (oral equivalent); OR C) A Gram-positive blood culture. If the Gram-positive isolate is S. aureus, it must be cultured from at least 1 culture bottle from either the peripheral set or the catheter set of culture bottles. For all other Gram-positive pathogens (eg, coagulase-negative staphylococci), isolates need to be cultured from at least 2 culture bottles of which one must be from the peripheral set. There must be no other obvious source of the bacteremia
* Presence of at least one of the following systemic signs of infection (may be obtained up to 24 hours prior to baseline): *Hypotension, defined as systolic blood pressure <90 mmHg or its reduction by >= 40 mmHg from the patient's baseline, in the absence of other causes for hypotension; *Tachycardia defined as a pulse rate > 90 beats per minute; *Tachypnea defined as a respiratory rate > 20 breaths per minute or PACO2 <32 torr; *White blood count >10,000 cells/mm3 or < 4,000 cells/mm3, or with a differential count showing >10% band neutrophil forms.
* Patients on hemodialysis with tunneled or nontunneled catheters including antibiotic coated hemodialysis catheters. Patients may have more than one concurrent catheter.
* Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* Patients presenting with any of the following will not be included in this study:
* Catheter-related bloodstream infections caused by Gram-negative bacteria, fungi, mixed cultures of Gram negative bacteria and Gram positive bacteria or mixed cultures of Gram positive/negative bacteria and fungi
* Patients with evidence of other infections resulting in bacteremia, such as clinical or radiographic signs of osteomyelitis, endocarditis, skin/skin structure infection, pneumonia, urinary tract infection, joint infection, intraabdominal infection, septic thrombophlebitis or other infection
* Patients in whom the infected catheter cannot be removed
* Patients with permanent intravascular devices such as artificial vascular grafts, implantable pacemakers or defibrillators; intra-aortic balloon pumps, and left ventricular assist device; intravascular transplants such as prosthetic cardiac valves; or non-intravascular devices such as peritoneal dialysis catheters; or neurosurgical devices such as ventriculo-peritoneal shunts, intra-cranial pressure monitors, or epidural catheters, prosthetic cardiac valves, prosthetic vascular grafts, or other internal prosthesis
* Females of child-bearing potential who are unable or unwilling to take adequate contraceptive precautions, have a positive pregnancy result within 24 hours prior to study entry, are known to be pregnant, or are currently breastfeeding an infant
* Identification of a pathogen resistant to linezolid or vancomycin
* Patients who are unlikely to survive through the treatment period and evaluation
* Administration of a glycopeptide antibiotic within 5 days prior to enrollment. Administration of other potentially effective systemic Gram-positive antibiotics for more than 48 hours within 72 hours prior to enrollment unless the pathogen showed drug resistance
* Previous enrollment in this protocol
* Hypersensitivity to linezolid, vancomycin, gentamicin or one of their excipients (or aztreonam if non-bacteremic Gram-negative coverage is required)
* Concurrent use of another investigational medication or use within 30 days of study entry
* Patients with pressor and fluid-resistant hemodynamic compromise or pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-09; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Pfizer Investigational Site, Baltimore, Maryland, United States
- Colombia (3):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Bogotá, D.C
- India (5):
  - Pfizer Investigational Site, Hyderbad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, New Delhi, National Capital Territory of Delhi
  - Pfizer Investigational Site, Chandigarh, Punjab
  - Pfizer Investigational Site, Chennai, Tamil Nadu
- Pfizer Investigational Site, Tel Aviv, Israel
- Pfizer Investigational Site, Imperia, Italy
- Pfizer Investigational Site, Częstochowa, Poland
- Slovakia (2):
  - Pfizer Investigational Site, Banská Bystrica, Slovakia
  - Pfizer Investigational Site, Nitra

REFERENCES:
- [Derived] Almeida BM, Moreno DH, Vasconcelos V, Cacione DG. Interventions for treating catheter-related bloodstream infections in people receiving maintenance haemodialysis. Cochrane Database Syst Rev. 2022 Apr 1;4(4):CD013554. doi: 10.1002/14651858.CD013554.pub2. PMID 35363884
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951105&StudyName=Linezolid%20in%20the%20Treatment%20of%20Hemodialysis%20Patients%20with%20Catheter-Related%20Gram-Positive%20Bloodstream%20Infections

RESULTS

PARTICIPANT FLOW:
Groups:
- Linezolid: Participants with catheter-related Gram-positive bloodstream infections received linezolid 600 milligram (mg) either intravenous injection or per oral tablet every 12 hours (hrs) along with intravenous gentamicin at a loading dose of 2 milligram/kilogram (mg/kg) body weight and subsequent doses targeted to keep serum peak levels between 6 to 8 microgram per milliliter (mcg/mL) and trough levels less than 1 mcg/mL, up to a maximum of 28 days.
- Vancomycin/Cefazolin: Participants with catheter-related Gram-positive bloodstream infections received vancomycin intravenously at a loading dose of 15 mg/kg body weight and subsequent doses targeted to keep serum trough levels between 10 to15 mcg/mL along with intravenous gentamicin at a loading dose of 2 mg/kg body weight and subsequent doses targeted to keep serum peak levels between 6 to 8 mcg/mL and trough levels less than 1 mcg/mL. Participants with a methicillin susceptible Gram-positive pathogen and not allergic to penicillin received cefazolin 1 gram (g) intravenously every 24 hours.
Period: Overall Study
Arm/Group | Linezolid | Vancomycin/Cefazolin
Started | 30 | 31
Completed | 9 | 14
Not Completed | 21 | 17
Not completed — Lack of Efficacy | 1 | 2
Not completed — Death | 3 | 0
Not completed — Adverse Event | 3 | 1
Not completed — Other | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linezolid | Vancomycin/Cefazolin | Total
Number analyzed (Participants) | 30 | 31 | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (17.7) | 49.7 (15.4) | 52.0 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Microbiological Response at Test-of-Cure (TOC) Visit
Description: Microbiological response assessed at participant level. Eradication = baseline isolate not present in repeat culture from the original infection site; Presumed Eradication = clinical response of cure based on Sponsor's (Sp) assessment, culture data not available for participants; Persistence = baseline isolate present in repeat culture from the original infection site; Presumed Persistence = culture data not available for participants with a clinical response of failure based on Sp assessment.
Time Frame: Short term follow-up (STFU) visit for TOC (2 to 3 weeks after the last dose of study medication)
Population: Data was not analyzed because there were not enough participants to perform a meaningful efficacy analysis due to early termination of the study.
Measure: Number; unit: participants
Arm/Group | Linezolid | Vancomycin/Cefazolin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Clinical Outcome Based on Sponsor's (Sp) and Investigator's (Ir) Assessment
Description: Ir assessment Cure: clinical signs/symptoms of infection (SSx) resolved and no reoccurrence; Improvement: Moderate resolution of SSx, no additional antibiotic needed; Failure: persistence/progression of baseline SSx, new clinical findings; Indeterminate: circumstances precluding above classification. Sp assessment Failure: concomitant antibiotic after day 3 up to/including Ir assessment day at TOC/upper limit of TOC window (if no Ir assessment at TOC), no Ir assessment at end of treatment (EOT) and TOC; Indeterminate: Sp assessment cured/ improved at EOT, no Ir assessment at TOC/indeterminate.
Time Frame: EOT (within 72 hours after last dose of study medication), STFU visit for TOC (2 to 3 weeks after the last dose of study medication), Long term follow-up (LTFU) visit (6 to 8 weeks after the last dose of study medication)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Linezolid | Vancomycin/Cefazolin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Complications During Therapy
Description: Late metastatic sequelae associated with Gram positive bacterial infections: abdominal abscess, brain abscess, meningitis, septic arthritis, osteomyelitis, endocarditis, empyema, spinal epidural abscess, intracerebral epidural abscess, septic phlebitis and septic thrombophlebitis.
Time Frame: LTFU visit (6 to 8 weeks after the last dose of study medication)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Linezolid | Vancomycin/Cefazolin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Pathogens Eradicated
Description: Eradication included Documented or Presumed Eradication of the given pathogen. Percentage of pathogen eradicated was calculated as number of pathogens eradicated divided by number of pathogens eradicated or persisted multiplied by 100.
Time Frame: STFU visit for TOC (2 to 3 weeks after the last dose of study medication), LTFU visit (6 to 8 weeks after the last dose of study medication)
Population: as for outcome 1
Measure: Number; unit: Percentage of Pathogens
Arm/Group | Linezolid | Vancomycin/Cefazolin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Eradication of Staphylococcus Aureus Nasal Colonization
Description: Eradication was defined as the absence of the original baseline nasal Staphylococcus aureus isolated in nasal swab culture.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin/Cefazolin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Linezolid | Vancomycin/Cefazolin
Serious Adverse Events (participants affected / at risk) | 7/30 | 3/31
Other Adverse Events (participants affected / at risk) | 12/30 | 9/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linezolid (N=30) | Vancomycin/Cefazolin (N=31)
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linezolid (N=30) | Vancomycin/Cefazolin (N=31)
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1
Asthenia (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 3
Candidiasis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Efficacy results were not reported because the study was prematurely terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.